CLINICAL TRIAL: NCT07127874
Title: First-in-Human, Phase 1 Study of PHN-012, an Antibody Drug Conjugate, in Patients With Advanced Solid Tumors
Brief Title: A Study of PHN-012 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pheon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PHN-012-001
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer; Pancreatic Cancer; Lung Cancer (NSCLC); Advanced Cancer; Advanced Solid Tumors
Keywords: Antibody Drug Conjugate; Carcinoma; Cancer; Solid Tumor
MeSH Terms: conditions — Colonic Neoplasms; Pancreatic Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1a and Phase 1b (Experimental): PHN-012 is administered intravenously
  Interventions: Drug: PHN-012

INTERVENTIONS:
Drug: PHN-012 — PHN-012 is an ADC

SUMMARY:
This first-in-human study will evaluate safety, tolerability, anti-tumor activity, immunogenicity, pharmacokinetics and pharmacodynamics of PHN-012, a novel antibody-drug conjugate (ADC), in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed, advanced/metastatic:

  1. Colorectal adenocarcinoma (CRC), or
  2. Non-small cell lung cancer (NSCLC), or
  3. Pancreatic ductal adenocarcinoma (PDAC).
* Has received at least one prior systemic therapy and radiologically or clinically determined progressive disease during or after the most recent line of therapy, and for whom no further standard therapy is available or who is intolerant to standard therapy.
* Has measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has adequate organ function.
* Has available tumor tissue sample at screening (either an archival specimen or fresh biopsy material).

Exclusion Criteria:

* Had prior treatment with any ADC containing topoisomerase-1 inhibiting payload.
* Has unstable central nervous system metastasis.
* Has persistent toxicities from previous systemic anti-cancer treatments of Grade >1.
* Has received systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the study drug.
* Has received wide-field radiotherapy (> 30% of marrow-bearing bones) within 28 days, or focal radiation for analgesic purpose or for lytic lesions at risk of fracture within 14 days prior to first dose of the study drug, or no recovery from side effects of such intervention.
* Had major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to first dose of the study drug, or no recovery from side effects of such intervention.
* Has a history of non-infectious pneumonitis (NIP) / interstitial lung disease (ILD) requiring systemic steroids within 6 months prior to first dose of the study drug, active NIP / ILD or suspected NIP / ILD which cannot be ruled out by imaging for Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (Phase 1a) | 12 months
Type, incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (Phase 1a) | 12 months
Frequency of dose interruptions, reductions, and discontinuations (Phase 1a and 1b) | 24 months
Overall response rate (ORR) (Phase 1b) | 12 months

SECONDARY OUTCOMES:
Best overall response (BOR) (Phase 1a and 1b) | 24 months
Disease control rate (DCR) (Phase 1a and 1b) | 24 months
Progression free survival (PFS) (Phase 1a and 1b) | 24 months
Time to response (TTR) (Phase 1a and 1b) | 24 months
Overall survival (OS) (Phase 1a and 1b) | 24 months
Pharmacokinetics, maximum concentration (Cmax) of total ADC (Phase 1a and 1b) | 24 months
Pharmacokinetics, Cmax of total antibody (Phase 1a and 1b) | 24 months
Pharmacokinetics, Cmax of free payload (Phase 1a and 1b) | 24 months
Pharmacokinetics, time of Cmax (Tmax) of total ADC (Phase 1a and 1b) | 24 months
Pharmacokinetics, Tmax of total antibody (Phase 1a and 1b) | 24 months
Pharmacokinetics, Tmax of free payload (Phase 1a and 1b) | 24 months
Pharmacokinetics, area under the curve (AUC) of total ADC (Phase 1a and 1b) | 24 months
Pharmacokinetics, AUC of total antibody (Phase 1a and 1b) | 24 months
Pharmacokinetics, AUC of total free payload (Phase 1a and 1b) | 24 months
Pharmacokinetics, terminal half-life (t1/2) of total ADC (Phase 1a and 1b) | 24 months
Pharmacokinetics, t1/2 of total antibody (Phase 1a and 1b) | 24 months
Pharmacokinetics, t1/2 of free payload (Phase 1a and 1b) | 24 months
Concentration of anti-drug antibodies (Phase 1a and 1b) | 24 months
Type, incidence and severity of AEs and SAEs (Phase 1b) | 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - PHN-012-001 Site, Washington D.C., District of Columbia
  - PHN-012-001 Site, Boston, Massachusetts
  - PHN-012-001 Site, Durham, North Carolina
  - PHN-012-001 Site, Nashville, Tennessee
  - PHN-012-001 Site, Houston, Texas
  - PHN-012-001 Site, San Antonio, Texas
  - PHN-012-001 Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No